CLINICAL TRIAL: NCT00786279
Title: Alcohol and Atherosclerosis Pilot Study
Acronym: AAAPILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kenneth Mukamal, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2008P-000164 AAAPILOT; R21AA016110 (NIH); 1R21AA016110 (NIH); NCT01377727 (obsolete NCT alias)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): 150 cc daily of flavored, calorie-free beverage without alcohol
  Interventions: Other: Ethanol-free beverage
- 2 (Experimental): 150 cc flavored, calorie-free beverage with 15 gm ethanol daily
  Interventions: Other: ethanol

INTERVENTIONS:
Other: ethanol — 15 gm ethanol daily for 6 months
  Arms: 2
Other: Ethanol-free beverage — 0 grams ethanol daily for 6 months.
  Arms: 1

SUMMARY:
We propose a pilot study to determine the feasibility of a long-term clinical trial of alcohol intake on atherosclerosis, the first step in determining whether moderate drinking prevents cardiovascular disease and hence in understanding the full health effects of alcohol across the population. We will randomize 40 participants aged 55 and older to a six-month period of consumption of 1 glass per day of either pure alcohol (diluted to the strength of wine) or water. At baseline and after 6 months, we will measure several standard and novel cardiovascular risk markers in the blood and will perform magnetic resonance imaging to measure atherosclerosis of the aorta.

DETAILED DESCRIPTION:
The feasibility of a long-term randomized trial of alcohol intake on clinical endpoints is uncertain. One approach that could minimize the size and duration of such a randomized trial would be to assess the effect of alcohol on progression of radiologically-defined atherosclerosis.

We propose a proof-of-principle pilot study of the effect of longer-term alcohol intake on atherosclerosis. We will recruit and randomize 40 participants aged 55 and older at high risk for CHD to a six-month period of consumption of a single 150 ml glass per day of either 10% ethanol (approximating wine) or water. At baseline and after 6 months, we will assess aortic atherosclerosis using magnetic resonance imaging. We will determine adherence in several ways, including serum markers, dietary recalls, and measurement of unused beverage. The primary outcomes in this feasibility study will be compliance with alcohol intake and the two MRI examinations. As secondary outcomes, we will measure standard and novel cardiovascular risk markers, including inflammatory markers and measures of glucose metabolism. We will assess safety on a continual basis, including repeated testing of liver enzymes and blood counts.

If successful, this pilot study will form the basis for a more definitive trial to determine the effect of alcohol intake on progression of atherosclerosis, which could itself establish the feasibility of even larger, longer-term studies of alcohol intake and occurrence of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Current Smoking
* Hypertension
* Family history of heart disease
* High LDL Cholesterol (>130 mg/dl)
* Low HDL CHolesterol (<40 mg/dl)
* Body Mass Index of 30 kg/m^2
* Waist circumference greater than 40 inches for men and 35 inches for women
* Report intake of at least one drink in the last month
* Post-menopause (if woman)

Exclusion Criteria:

* History of myocardial infarction (MI)/ heart attack within prior 6 months.
* Revascularization procedure (coronary, carotid, or peripheral)
* Stroke
* Claustrophobia
* Intolerance to previous MRI examinations
* Standard MRI contraindications (e.g. pacemaker, intra-auricular implants, or intracranial clips)
* Weight over 350 pounds
* Active atrial fibrillation
* Reports intake of more than 7 drinks per week currently, has previous or current history of alcohol abuse based on standard questionnaires, or who has consumed more than 4 drinks in one day within the last 6 months.
* Intolerance or allergy to alcohol consumption (includes flushing)
* Allergy to aspartame, acesulfame, or artificial food coloring
* Any severe illness expected to cause death or profound disability within 6 months
* Evidence of depression (as measured based on a Center for Epidemiological Studies Depression score of 16 or higher)
* History of chronic liver disease
* Personal history of breast or any gastrointestinal cancer, uncontrolled hypertension (blood pressure greater than or equal to 180/110)
* Chronic renal failure on dialysis
* Current use of Metronidazole or Warfarin
* Use of benzodiazepines, barbiturates, and related sedative/ hypnotics 4 or more days per week.
* Severe psychiatric illness
* Inability to speak English
* Lack of a working telephone

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Adherence to alcohol intake and MRI examinations | 6 months

SECONDARY OUTCOMES:
GGT | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Mukamal, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Panagiotou G, Mu L, Na B, Mukamal KJ, Mantzoros CS. Circulating irisin, omentin-1, and lipoprotein subparticles in adults at higher cardiovascular risk. Metabolism. 2014 Oct;63(10):1265-71. doi: 10.1016/j.metabol.2014.06.001. Epub 2014 Jun 9. PMID 25060690
- [Derived] Mukamal KJ, Na B, Mu L, Mantzoros CS, Manning WJ, Mittleman MA. Lessons and Challenges from a 6-Month Randomized Pilot Study of Daily Ethanol Consumption: Research Methodology and Study Design. Curr Dev Nutr. 2017 Jun 15;1(7):e000505. doi: 10.3945/cdn.117.000505. eCollection 2017 Jul. PMID 29955710